CLINICAL TRIAL: NCT02575573
Title: Influencing Factors on Resuscitation Decisions in the ED
Brief Title: Resuscitation Decisions in the Emergency Department (ED)
Acronym: REDEED
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Max Planck Institute for Human Development (Other)
Responsible Party: Sponsor
Other Study IDs: REDEED
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Resuscitation
Keywords: resuscitation decision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Admitted patients at the ED
  Interventions: Other: Factors influencing resuscitation decisions of patients; Other: Factors leading to not asking patients about resuscitation preference

INTERVENTIONS:
Other: Factors influencing resuscitation decisions of patients
Other: Factors leading to not asking patients about resuscitation preference

SUMMARY:
The investigators will retrospectively examine the connection between resuscitation decisions of admitted patients at the ED of the University Hospital of Basel and several demographic and health related measures. Additionally there will be an examination, which patient characterestics may have lead to patients not having been asked about resuscitation decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department (duration of hospitalisation more than 24 h).
* Patients with a research consent "yes".

Exclusion Criteria:

* Patients being discharged within less than 24 hours.
* Patients with a research consent "no".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients from the Emergency Department of the University Hospital of Basel between the 1st of January 2010 and the 31st of December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Resuscitation decision of the patient | During stay at ED (range: <1 hour until 31 days)
  Answer to the question "Do you want life prolonging treatment if necessary?"

SECONDARY OUTCOMES:
Patient characterestics, which may have lead to patients not having been asked about resuscitation decisions | During stay at ED (range: <1 hour until 31 days)
  Age, gender, resuscitation decision, ICD codes

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, Prof., Principal Investigator — University Hospital Basel, Emergency Department
Locations (1):
- University Hospital Basel, Emergency Department, Basel, Canton of Basel-City, Switzerland